CLINICAL TRIAL: NCT04589416
Title: Erciyes University Clinical Research Ethics Committee
Brief Title: Clinical Evaluation Of Class I Composite Resin Restorations Using Three Different Adhesive Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Nazire Nurdan Çakır, Assist. Prof Nazire Nurdan Çakır, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 5930
Record Dates: First submitted 2020-10-03; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dental Adhesive Materials
Keywords: Adhesive system; Clinical follow-up; Class I restoration; Composite resin; FDI; USPHS

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Bond 2 (Active Comparator): Single Bond 2 is a traditional etch and rinse adhesive system. It is used to bond the composite resin to the dental tissues. It was applied to the cavities opened in accordance with the manufacturer's instructions.
  Interventions: Other: Dental adhesive materials.
- Clearfil SE Bond (Active Comparator): Clearfil SE bond is traditional two step self-etch adhesive system. It is used to bond the composite resin to the dental tissues. It was applied to the cavities opened in accordance with the manufacturer's instructions.
  Interventions: Other: Dental adhesive materials.
- Tri-S Bond (Active Comparator): Tri-S bond is traditional one step self-etch adhesive system. It is used to bond the composite resin to the dental tissues. It was applied to the cavities opened in accordance with the manufacturer's instructions.
  Interventions: Other: Dental adhesive materials.

INTERVENTIONS:
Other: Dental adhesive materials. — It is used to bond the composite resin to the dental tissues. That is, it is used to bond dental filling materials to dental tissues.

SUMMARY:
Nowadays, most composite resins require the use of an adhesive material prior to application. For this purpose, etch & rinse (ER) and self-etch (SE) systems have been used for many years. While many in-vitro studies have been conducted in the literature comparing three adhesive systems, the number of clinical studies is less and inadequate. Therefore, the aim of this study was to investigate the effect of 3 different adhesive systems commonly used in clinics on the success of class I composite restorations using the criteria of the World Dental Federation (FDI) and the United States Public Health Service (USPHS).

DETAILED DESCRIPTION:
Nowadays, most composite resins require the use of an adhesive material prior to application. For this purpose, etch & rinse (ER) and self-etch (SE) systems have been used for many years. Compared to SE systems, which are simplified and very easy to use, requiring less technical precision, traditional ER systems are still very popular and preferred by dentists. However, current researchers indicate that ER systems are more effective on enamel than dentin and that this effect is better than SE systems. SE systems are approaches in which the acid application and washing step are eliminated clinically and the possibility of making mistakes during the application and manipulation is reduced. An important advantage of these systems is that demineralization and resin infiltration occurs at the same time. Clinically, the application times are shorter than traditional systems. Two-steps SE systems have been used for a long time. In this system, the need for a separate acidic primer application has needed clinicians reason to search for single-steps bonding agents. And, in recent years, single-step SE systems also called "all in one", have been developed that include all steps of pickling, primer application, and adhesive agent application. However, there are studies showing that these systems do not perform as well as two-step SE systems. While many in-vitro studies have been conducted in the literature comparing three adhesive systems, the number of clinical studies is less and inadequate. Therefore, the aim of this study was to investigate the effect of 3 different adhesive systems commonly used in clinics on the success of class I composite restorations using the criteria of the World Dental Federation (FDI) and the United States Public Health Service (USPHS).

ELIGIBILITY:
Inclusion Criteria:

* At least 3 Class-I caries lesions
* Good health
* Acceptable level of oral hygiene

Exclusion Criteria:

* Did not have four caries lesions at least
* Did not have Class-II caries lesions
* Deep caries reaching the pulp
* The patients are not 18-22 years old
* Bruxism
* Periodontal disease
* Refused to participate

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation Of Class I Composite Resin Restorations Using Three Different Adhesive Systems with FDI and USPHS criteria | One years
  FDI; World Dental Federation USPHS; United States Public Health Service. Two calibrated observers who were blinded to the objective of this study performed the evaluations.
Clinical Evaluation Of Class I Composite Resin Restorations Using Three Different Adhesive Systems with FDI and USPHS criteria | Two years
  FDI; World Dental Federation USPHS; United States Public Health Service. Two calibrated observers who were blinded to the objective of this study performed the evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Nazire Nurdan Çakır, Principal Investigator — Nuh Naci Yazgan University

IPD SHARING:
Plan to Share IPD: Undecided